CLINICAL TRIAL: NCT02583386
Title: Comprehensive Fall Prevention and Detection in Multiple Sclerosis
Acronym: FFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portland VA Medical Center (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Michelle H. Cameron, MD, PT, MCR, Neurologist, Portland VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3516
Record Dates: First submitted 2015-10-19; First posted 2015-10-22 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2020-03

CONDITIONS: Multiple Sclerosis
Keywords: mobility; falls; fall prevention; gait and balance; automatic fall detector
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Free From Falls training group (Active Comparator): Subjects randomized to this group will receive an 8 week exercise and educational program on fall prevention (Free From Falls fall prevention program). They will have mobility and quality of life assessments taken at baseline, after the training program has been completed, and 3 and 6 months later. During this time, their falls will be recorded monthly using prospective falls calendars.
  Interventions: Behavioral: Free From Falls fall prevention program
- Wait-list control group (No Intervention): Subjects in this group will participate in the same mobility and quality of life assessments and completion of the falls calendars, but will receive no training classes during this time. These subjects will have the opportunity to receive the class sessions when all assessment visits have been completed.
- FFF training group w/ Fall Detector (Active Comparator): Subjects randomized to this group will receive an 8 week exercise and educational program on fall prevention (Free From Falls fall prevention program). They will have mobility and quality of life assessments taken at baseline, after the training program has been completed, and 3 and 6 months later. During this time, their falls will be recorded monthly using prospective falls calendars.
  In addition, this group will be asked to wear electronic fall detectors on their bodies for the first 10 weeks of their participation in the study.
  Interventions: Behavioral: Free From Falls fall prevention program; Other: Electronic Fall Detector
- Wait-list control w/ Fall Detector (Other): Subjects in this group will participate in the same mobility and quality of life assessments and completion of the falls calendars, but will receive no training classes during this time. These subjects will have the opportunity to receive the class sessions when all assessment visits have been completed.
  In addition, this group will be asked to wear electronic fall detectors on their bodies for the first 10 weeks of their participation in the study.
  Interventions: Other: Electronic Fall Detector

INTERVENTIONS:
Behavioral: Free From Falls fall prevention program — Eight-week education and exercise program, intended to reduce falls in people with Multiple Sclerosis.
  Arms: FFF training group w/ Fall Detector; Free From Falls training group
Other: Electronic Fall Detector — 30 participants will be randomly selected to wear an electronic fall detector during the first 10 weeks of study participation. This fall detector will automatically record any falls occurring while worn.
  Arms: FFF training group w/ Fall Detector; Wait-list control w/ Fall Detector

SUMMARY:
The purpose of this study is to examine whether an exercise and educational classroom program can help reduce falls in people with Multiple Sclerosis who fall frequently.

DETAILED DESCRIPTION:
The investigators will recruit 94 people with Multiple Sclerosis, who report having fallen at least twice in the previous 2 months. Participants will be randomized to be placed in either a group that receives classroom training during the study, or into a wait-listed control group that will be offered the classroom training after their participation in the study is completed. All participants will receive mobility and quality of life assessments at baseline, 9 weeks, 5 months, and 8 months. All participants will be asked to record any falls they have on falls calendars.

In addition, 30 participants will be randomized to wear electronic fall detectors on their bodies for the duration of the study. These detectors will record when and where falls occur, and this data will be compared with the participants' self-reported falls as recorded on the falls calendars.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis of any type,
* self-reported history of 2 or more falls in the previous 2 months,
* Expanded Disability Status Scale of ≤ 6.0 (i.e. able to walk at least 100 meters with or without a walking aid),
* be willing and intellectually able to understand and to sign an informed consent, and to adhere to protocol requirements,
* have sufficient motor function to complete a written daily record of falls for 8 months,
* be community dwelling.

Exclusion Criteria:

* have a self-reported musculoskeletal or neurological condition other than MS that is known to affect balance or gait and is associated with falls, such as a lower-extremity joint replacement within the past year, peripheral neuropathy, vestibular disorder, alcoholism, stroke, or seizures.
* be unable to follow directions in English,
* have unhealed bone fractures or other condition that may put them at risk of injury during balance training and assessments,
* blind (visual acuity corrected worse than 20/200),
* serious psychiatric or medical conditions that would preclude reliable participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-04; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Self-Reported Falls and Fall-Related Injuries at Completion of Program and the Following Six Months | At baseline, at program completion (9 weeks), 3 months after program completion (9 weeks + 3 months), 6 months after program completion (9 weeks + 6 months)
  Paper fall calendars
Change from Baseline in Balance Confidence | At baseline, at program completion (9 weeks), 3 months after program completion (9 weeks + 3 months), 6 months after program completion (9 weeks + 6 months)
  Activities-specific Balance Confidence questionnaire
Change from Baseline in Satisfaction with Participation in Social Roles | At baseline, at program completion (9 weeks), 3 months after program completion (9 weeks + 3 months), 6 months after program completion (9 weeks + 6 months)
  Patient Reported Outcomes Measurement Information System (PROMIS) Item Bank v. 1.0 - Satisfaction with Participation in Social Roles
Change from Baseline in Ability to Participate in Social Roles and Activities | At baseline, at program completion (9 weeks), 3 months after program completion (9 weeks + 3 months), 6 months after program completion (9 weeks + 6 months)
  Patient Reported Outcomes Measurement Information System (PROMIS) Item Bank v. 2.0 - Ability to Participate in Social Roles and Activities
Change from Baseline in Quality of Life | At baseline, at program completion (9 weeks), 3 months after program completion (9 weeks + 3 months), 6 months after program completion (9 weeks + 6 months)
  Multiple Sclerosis Impact Scale-29
Accuracy and Impact of Fall Detection and Localization by the MobileRF Fall Detection System, Compared to Paper Fall Calendars | 8 weeks
  The Mobile RF Fall Detection System automatically records falls per day experienced by the wearer. The results obtained by the fall detector will be tested for accuracy against the self-reported falls reported on paper fall calendars, in which participants manually record falls per day on a paper log.

SECONDARY OUTCOMES:
Change from Baseline in Mobility and Balance (TUG score) at Completion of Program and the Following Six Months | At baseline, at program completion (9 weeks), 3 months after program completion (9 weeks + 3 months), 6 months after program completion (9 weeks + 6 months)
  Timed Up and Go
Change from Baseline in Mobility and Balance (FSST score) at Completion of Program and the Following Six Months | At baseline, at program completion (9 weeks), 3 months after program completion (9 weeks + 3 months), 6 months after program completion (9 weeks + 6 months)
  Four Square Step Test
Change from Baseline in Level of Physical Activity at Completion of Program and the Following Six Months | At baseline, at program completion (9 weeks), 3 months after program completion (9 weeks + 3 months from baseline), 6 months after program completion (9 weeks + 6 months + baseline)
  International Physical Activity Questionnaire, short form
Change from Baseline in Fall Prevention Strategy at Completion of Program and the Following Six Months | At baseline, at program completion (9 weeks), 3 months after program completion (9 weeks + 3 months), 6 months after program completion (9 weeks + 6 months)
  Fall Prevention Strategy Survey
Change from Baseline in Fatigue at Completion of Program and the Following Six Months | At baseline, at program completion (9 weeks), 3 months after program completion (9 weeks + 3 months), 6 months after program completion (9 weeks + 6 months)
  Patient Reported Outcomes Measurement Information System (PROMIS) Item Bank v. 1.0 - Fatigue
Change from Baseline in Mobility at Completion of Program and the Following Six Months | At baseline, at program completion (9 weeks), 3 months after program completion (9 weeks + 3 months), 6 months after program completion (9 weeks + 6 months)
  Patient Reported Outcomes Measurement Information System (PROMIS) Item Bank v. 1.2 - Physical Function - Mobility
Change from Baseline in Psychosocial Function at Completion of Program and the Following Six Months | At baseline, at program completion (9 weeks), 3 months after program completion (9 weeks + 3 months), 6 months after program completion (9 weeks + 6 months)
  Patient Reported Outcomes Measurement Information System (PROMIS) Item Bank v. 1.0 - Psychosocial Illness Impact - Positive
Change from Baseline in Knowledge and Confidence Regarding Fall Prevention at Completion of Program and the Following Six Months | At baseline, at program completion (9 weeks), 3 months after program completion (9 weeks + 3 months), 6 months after program completion (9 weeks + 6 months)
  Fall Prevention Knowledge and Confidence Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michelle H. Cameron, MD, PT, MCR, Principal Investigator — Portland VA Medical Center
Locations (1):
- VA Portland Health Care System, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hildebrand A, Jacobs PG, Folsom JG, Mosquera-Lopez C, Wan E, Cameron MH. Comparing fall detection methods in people with multiple sclerosis: A prospective observational cohort study. Mult Scler Relat Disord. 2021 Nov;56:103270. doi: 10.1016/j.msard.2021.103270. Epub 2021 Sep 20. PMID 34562766